CLINICAL TRIAL: NCT07407881
Title: Effectiveness of Manual Pressure Application Versus Shotblocker on Reducing Insulin Injection Pain Among Children With Type 1 Diabetes Mellitus
Brief Title: Shot Blocker and Manual Pressure Application
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Shotblocker and manual pressur
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Injection Pain Prevention
Keywords: Manual pressure and shotblocker

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Manual Pressure (Experimental): Manual Pressure Application (MPA) is a cost-free, nonpharmacological method that is easily learned and requires no equipment or preparation use for reduce insulin injection pain among children with type 1 diabetes mellitus .Manual therapy interventions (also described as force-based manipulations) refer to the passive application of mechanical force to the outside of the body with therapeutic effect. Right thumb pressure was be applied to the appropriate inject site of insulin therapy for 10 seconds, then immediately inject the insulin. The children's pain intensity during and immediately after insulin injection scores will be rated by the children themselves and a researcher using the Wong-Baker FACES Pain Rating Scale.
  Interventions: Other: Manual pressure applied at injection site during insulin injection to reduce pain
- Arm 2 : shotblocker (Experimental): The Shotblocker is a low-technology, cost-effective small flat C-shaped plastic flexible tool with multiple short, blunt protrusions on one side that is a non-invasive and drug-free method. This tool is applied to the skin to create signal sensory distraction surrounding the injection site, resulting in inhibition of pain signals during injection. Apply the shotblocker and press firmly with its multiple blunt protrusions on contact points of skin. After that, give an insulin injection through the central opening. The children's pain intensity during and immediately after insulin injection scores will be rated by the children themselves and a researcher using the Wong-Baker FACES Pain Rating Scale.
  Interventions: Device: Shotblocker
- Arm 3: Control group (Active Comparator): The children's pain intensity scores during and immediately after insulin injection will be rated by the children themselves and a researcher by using the Wong-Baker FACES Pain Rating Scale to control the group who don't receive the previous method of intervention and receive routine care only.
  Interventions: Other: Control group stander care

INTERVENTIONS:
Other: Manual pressure applied at injection site during insulin injection to reduce pain — Right thumb pressure was be applied to the appropriate inject site of insulin therapy for 10 seconds, then immediately inject the insulin. The children's pain intensity during and immediately after insulin injection scores will be rated by the children themselves and a researcher using the Wong-Baker FACES Pain Rating Scale.
  Other Names: Manual pressure technique
  Arms: Arm 1: Manual Pressure
Device: Shotblocker — Apply the shotblocker and press firmly with its multiple blunt protrusions on contact points of skin. After that, give an insulin injection through the central opening. The children's pain intensity during and immediately after insulin injection scores will be rated by the children themselves and a researcher using the Wong-Baker FACES Pain Rating Scale.
  Arms: Arm 2 : shotblocker
Other: Control group stander care — The children's pain intensity scores during and immediately after insulin injection will be rated by the children themselves and a researcher by using the Wong-Baker FACES Pain Rating Scale to control the group who don't receive the previous method of intervention and receive routine care only.
  Arms: Arm 3: Control group

SUMMARY:
Aim of my intervention to test the effectiveness of using the manual pressure application and shotblocker for relief insulin injection pain in children with type 1 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Their age ranging between 6 to12 years old of both genders. Diagnosed with Type 1 Diabetes Mellitus (new and old diagnosed). Receiving subcutaneous insulin injection .

Exclusion Criteria:

* Having lipodystrophy, infection and nerve damage at injection site. Tooking analgesic within the least 6 hours. Refusing to participate.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | during and immediately after insulin injection
  The children's pain intensity during and immediately after insulin injection scores will be rated by the children themselves and a researcher using the Wong-Baker FACES Pain Rating Scale.
Pain Intensity | Immediately after insulin injection
  The children's pain intensity during and immediately after insulin injection scores will be rated by the children themselves and a researcher using the Wong-Baker FACES Pain Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Fawzia El-Sayed Abusaad, Professor of pediatric Nursing, Study Director — Faculty of Nursing - Mansoura University
Locations (1):
- Mansura University Children's Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy considerations, and because no informed consent was obtained for data sharing beyond the objectives of this study.

REFERENCES:
- [Background] EL-mahdy, E. S. R., El-khedr, S. M., Elrifaey, S. M., & Elaraby, M. E. (2023). Effect of Shot Blockers versus Buzzy Bee Distractor on Relieving Pain and Anxiety Level during Insulin Injection among Children with Type I Diabetes. Tanta Scientific Nursing Journal, 29(2), 32-49. https://doi.org/10.21608/tsnj.2023.298374
- [Background] İyi Z, İşler A, Özer Z. Effectiveness of ShotBlocker application on reducing the pain of needle-related procedures in children: A systematic review and meta-analysis. J Pediatr Nurs. 2024 Sep-Oct;78:e438-e447. doi: 10.1016/j.pedn.2024.08.006. Epub 2024 Aug 10. PMID: 39129083.